CLINICAL TRIAL: NCT05073484
Title: A Phase 1, Multi-Center, Open-Label Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT6021 as Mono Therapy or in Combination With BAT1308 in Patients With Advanced Solid Tumors
Brief Title: Assessment of Safety and Preliminary Efficacy With BAT6021 in Solid Tumor Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the disclosed global research data on the same target drugs, the company has carefully considered and decided to terminate the project to optimize the existing research pipeline.
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-6021-002-CR
Record Dates: First submitted 2021-09-09; First posted 2021-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- 10 mg of BAT6021 (Experimental): BAT6021 100mg/vial，10mg Ⅳ infusions
  Interventions: Drug: BAT6021
- 30 mg of BAT6021 (Experimental): BAT6021 100mg/vial，30mg Ⅳ infusions
  Interventions: Drug: BAT6021
- 100 mg of BAT6021 (Experimental): BAT6021 100mg/vial，100mg Ⅳ infusions
  Interventions: Drug: BAT6021
- 300 mg of BAT6021 (Experimental): BAT6021 100mg/vial，300mg Ⅳ infusions
  Interventions: Drug: BAT6021
- 600 mg of BAT6021 (Experimental): BAT6021 100mg/vial，600mg Ⅳ infusions
  Interventions: Drug: BAT6021
- 900 mg of BAT6021 (Experimental): BAT6021 100mg/vial，900mg Ⅳ infusions
  Interventions: Drug: BAT6021
- 100mg BAT6021+300mg BAT1308 (Experimental): BAT6021 100mg/vial，BAT1308 100mg/vial ; BAT6021 100mg+BAT1308 300mg Ⅳ infusions
  Interventions: Drug: BAT6021; Drug: BAT1308
- 300mg BAT6021+300mg BAT1308 (Experimental): BAT6021 100mg/vial，BAT1308 100mg/vial ; BAT6021 300mg+BAT1308 300mg Ⅳ infusions
  Interventions: Drug: BAT6021; Drug: BAT1308
- 600mg BAT6021+300mg BAT1308 (Experimental): BAT6021 100mg/vial，BAT1308 100mg/vial ; BAT6021 600mg+BAT1308 300mg Ⅳ infusions
  Interventions: Drug: BAT6021; Drug: BAT1308

INTERVENTIONS:
Drug: BAT6021 — Ⅳ infusions
  Other Names: Recombinant Humanized Anti-TIGIT Antibody Solution for Injection
Drug: BAT1308 — Ⅳ infusions
  Other Names: Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection
  Arms: 100mg BAT6021+300mg BAT1308; 300mg BAT6021+300mg BAT1308; 600mg BAT6021+300mg BAT1308

SUMMARY:
This first-in-human open-label, multi center, dose-escalation and expansion study is designed to evaluate the safety, tolerability, and PK of BAT6021 alone or in combination with BAT1308 (an anti-PD-1 antibody) in participants with locally advanced, recurrent, or metastatic incurable tumors for whom standard therapy does not exist, has proven to be ineffective or intolerable, or is considered inappropriate, or for whom a clinical trial of an investigational agent is a recognized standard of care.

DETAILED DESCRIPTION:
Anti-PD-1 and anti-PD-L1 antibodies targeting the immuno-inhibitory PD-1 pathway (thus activating T cells) have achieved clinical success in many types of cancers. However, studies have shown that anti-TIGIT antibodies not only trigger T cells and Natural Killer(NK) cells, but they can also activate T cells to a greater extent than anti-PD-1 antibodies. Therefore, further clinical investigation of anti-TIGIT antibodies such as BAT6021 is warranted.

PD-1 and TIGIT are commonly co-expressed in T cells of the same tumor; thus, combining anti-TIGIT antibodies with PD-1/PD-L1 inhibitors may be a more effective cancer treatment. Indeed, anti-TIGIT antibodies have demonstrated synergy with anti-PD-1/PD-L1 antibodies in preclinical models. In addition, sponsor have shown that single administration of BAT1308 or BAT6021 could not effectively inhibit CT26 tumor growth in PD-1/TIGIT- humanized syngeneic mice; however, the combination treatment resulted in potent anti-tumor activity. Therefore, combined treatment with BAT6021 and an anti-PD-1/PD-L1 antibody like BAT1308 could improve therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give voluntary informed consent and understand the study and are willing to follow and complete all the test procedures.
2. Aged ≥ 18 years.
3. Life expectancy ≥ 3 months.
4. ECOG performance status ≤ 1.
5. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors that are refractory to standard therapy, or for whom no standard therapy exists.
6. Has measurable disease per RECIST v1.1. that was not in a prior radiation or other locally treated area, unless imaging-based progression has been clearly documented following radiation or other local therapy.

Exclusion Criteria:

1. Females who are pregnant or nursing.
2. Receiving concurrent anticancer therapy or investigational therapy (including chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy).
3. Has remaining AEs > Grade 1 from prior antitumor treatment as per CTCAE v5.0, with the exception of alopecia.
4. Participants with primacy central nervous system (CNS) malignancy, symptomatic CNS metastases, meningeal metastases or leptomeningeal disease are not allowed. Note: Participants with asymptomatic CNS metastases are eligible if clinically controlled, which is defined as 1) ≥ 4 weeks of stable neurologic function following CNS-directed therapy prior to Screening, 2) no evidence of CNS disease progression as determined by radiographic imaging ≥ 4 weeks prior to Screening, 3) ≥ 2 weeks from discontinuation of anti-seizure and steroid therapies (receiving prednisone ≤ 10mg or equivalent steroid therapies is allowed) prior to Screening.
5. Had major surgery within 28-days of the Screening Visit. Note: Participants who have undergone a non-major surgical procedure ≥ 28 days prior to Screening must have recovered adequately from the toxicity and/or complications from the intervention before administration of the first dose of study drugs.
6. History of tissue or organ transplantation.
7. History of severe infection deemed clinically significant by the PI or designee within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose of study drugs.
8. History of human immunodeficiency virus (HIV) infection or history of autoimmune diseases.
9. Active hepatitis B or C. Note: Hepatitis B virus (HBV) carriers without active disease (HBV DNA titer < 1000 copies/mL or 200 IU/mL) or cured Hepatitis C (negative HCV RNA test) may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | A minimum of 21 days after first dose of BAT6021
  DLT is defined as one of the following as investigator related to study drug:
  Grade 5 toxicity; Hematologic Toxicity ; ≥ Grade 4 anemia; Grade 4 thrombocytopenia that lasts for ≥ 7 days or Grade 3 thrombocytopenia, if associated with clinically significant bleeding (≥ Grade 2 hemorrhage) or requires transfusion of platelets; Grade 4 neutropenia that lasts for ≥ 7 days, or Grade 3 neutropenia that lasts for ≥ 7 days or with documented infection; Grade 3 or Grade 4 febrile neutropenia of any duration.
Serious adverse event（SAE） | From the time of informed consent to 90 days after the last dose or until the initiation of a new cancer treatment.
  Any SAE that is judged by the PI or designee to be related to the study medication must be reported regardless of the amount of time since the last dose received. Follow-up information collected for any initial report of an SAE must also be reported to the Sponsor (or its designee) within 24 hours of receipt by the PI or designee.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | every cycle until cycle 6 (one cycle equals 3 weeks)
  Cmax
Immunogenicity | every cycle until cycle 6 (one cycle equals 3 weeks)
  Presence of ADAs / neutralizing antibodies (NAbs).

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Pal, M.D, Ph.D, Principal Investigator — Medical Oncologist at cancer Therapy, Liverpool Hospital
Locations (3):
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - Cabrini Hospital Malvern, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD